CLINICAL TRIAL: NCT03897075
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Assess the Efficacy and Safety of Tildrakizumab in the Treatment of Moderate to Severe Nail Psoriasis
Brief Title: Efficacy and Safety Study of Tildrakizumab in the Treatment of Nail Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TILD-18-19
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Nail Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Tildrakizumab
- Arm B (Placebo Comparator)
  Interventions: Drug: Tildrakizumab; Drug: Placebo

INTERVENTIONS:
Drug: Tildrakizumab — PART 1: Double-blind Placebo-controlled PART 2: Double-blind Active Treatment Extension PART 3: Observational Safety Follow-up
Drug: Placebo — PART 1: Double-blind Placebo-controlled PART 2: Double-blind Active Treatment Extension PART 3: Observational Safety Follow-up
  Arms: Arm B

SUMMARY:
Phase 3b study to Assess the Efficacy and Safety of Tildrakizumab in the Treatment of Moderate to Severe Nail Psoriasis

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Subjects with a chronic moderate to severe plaque-type psoriasis for at least 6 months (as determined by subject interview and confirmation of diagnosis through physical examination by Investigator).
2. Subjects must have moderate to severe nail psoriasis at Screening and Baseline, defined by:

   * mNAPSI score of ≥20.
   * ViSENPsO ≥3
3. Subjects must have moderate to severe plaque psoriasis at Screening and Baseline, defined by:

   * s-PGA score of at least 3.
   * Body Surface Area (BSA) involvement of ≥10%.
   * PASI ≥12
4. Subjects must be considered candidates for systemic therapy, meaning psoriasis inadequately controlled by topical treatments (corticosteroids), and/or phototherapy, and/or previous systemic therapy.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. Subjects who have predominantly non-plaque forms of psoriasis, specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced, or medication-exacerbated psoriasis, or new-onset guttate psoriasis.
2. Subjects with ongoing inflammatory skin diseases other than psoriasis or any other disease affecting the fingernails, which may potentially confound the evaluation of study treatment.
3. Subjects with fungal nail infection should be excluded from the study. Subjects in whom the Investigator suspects a fungal nail infection in addition to nail psoriasis should have scrapings sent for direct microscopy and fungal culture. If fungal culture or direct microscopy of nail scrapings turns out to be positive for fungal infection, the subject should be excluded from the study. At the discretion of the investigator, Periodic Acid-Schiff (PAS) staining for nail clippings could also be considered to rule of fungal infection of the nails. Direct microscopy or fungal culture are not required if fungal infection is diagnosed in PAS staining.
4. Subjects with any previous use of tildrakizumab or other IL-23/Th-17 pathway inhibitors, including p40, p19 and IL-17 antagonists for psoriasis.
5. Subjects with known history of allergy or hypersensitivity to any of the inactive ingredients of the Tildrakizumab or placebo formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - California Dermatology & CRI (Site 18), Encinitas, California
  - First OC Dermatology (Site 07), Fountain Valley, California
  - Dermatology Research Associates (Site 09), Los Angeles, California
  - Clinical Science Institute (Site 14), Santa Monica, California
  - Florida Academic Centers Research and Education, LLC (Site 21), Coral Gables, Florida
  - Renstar Medical Research (Site 23), Ocala, Florida
  - Forest Hills Dermatology Group (Site 04), Forest Hills, New York
  - Clinical Partners, LLC (Site 08), Johnston, Rhode Island
  - Center for Clinical Studies Cypress (Site 17), Cypress, Texas
  - Center for Clinical Studies (Site 11), Houston, Texas
  - Progressive Clinical Research (Site 27), San Antonio, Texas
- Australia (6):
  - Premier Dermatology (Site 47), Kogarah, New South Wales
  - St George Dermatology & Skin Cancer Centre (Site 45), Kogarah, New South Wales
  - Veracity Clinical Research/ Specialist Connect(Site 44), Woolloongabba, QSLD
  - North Eastern Health Specialists (Site 46), Campbelltown, South Australia
  - Skin Health Institute Inc. (Site 43), Carlton, Victoria
  - Fremantle Dermatology (Site 40), Fremantle, WAUS

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects received placebo up to Week 28
- Tildrakizumab 100 mg: Subjects received Tildrakizumab 100 mg upto week 16.
Period: Overall Study
Arm/Group | Placebo | Tildrakizumab 100 mg
Started | 48 | 51
Completed | 35 | 43
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tildrakizumab 100 mg | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (15.14) | 46.6 (11.74) | 46.4 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 32 | 38 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 18 | 38
  Not Hispanic or Latino | 28 | 33 | 61
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieve at Least a 75% Improvement From Baseline in Total mNAPSI at Week 28.
Description: Primary Efficacy Endpoint
Time Frame: Week 28
Measure: Number; unit: proportion of subjects
Groups:
- Tildrakizumab 100 mg: Subjects received Tildrakizumab 100 mg up to week 16
Arm/Group | Placebo | Tildrakizumab 100 mg
Number analyzed (Participants) | 48 | 51
proportion of subjects | 0.042 | 0.255
Statistical Analysis 1: Comparison: Placebo vs Tildrakizumab 100 mg; Test type: Superiority; p = 0.00311, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Proportion of Subjects With a Score of "0 - Normal" or "1 - Minimal Nail Psoriasis" and at Least a 2-point Decrease From Baseline at Week 28 as Measured by the ViSENPsO.
Time Frame: Week 28
Measure: Number; unit: Proportion of subjects
Arm/Group | Placebo | Tildrakizumab 100 mg
Number analyzed (Participants) | 48 | 51
Proportion of subjects | 0.042 | 0.294
Statistical Analysis 1: Comparison: Placebo vs Tildrakizumab 100 mg; Test type: Superiority; p = 0.00079, Cochran-Mantel-Haenszel

3. Secondary Outcome: The Proportion of Subjects With at Least 3 Point Decrease From Baseline, in Nail Pain NRS Score in Subjects With Baseline Nail Pain NRS Score of >3
Time Frame: Week 28
Population: The number of subjects analysed represents the Intent-to-Treat population with baseline nail pain NRS ≥ 3
Measure: Number; unit: proportion of subjects
Arm/Group | Placebo | Tildrakizumab 100 mg
Number analyzed (Participants) | 35 | 33
proportion of subjects | 0.257 | 0.455
Statistical Analysis 1: Comparison: Placebo vs Tildrakizumab 100 mg; Test type: Superiority; p = 0.09892, Cochran-Mantel-Haenszel

4. Other Pre Specified Outcome: The Percentage of Subjects With Incidence, Seriousness, and Severity of All Adverse Events.
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

5. Other Pre Specified Outcome: The Percentage of Subjects With Severe Infections Whether or Not Reported as a Serious Event Defined as Any Infection Meeting the Regulatory Definition of a Serious Adverse Event, or Any Infection Requiring Intravenous Antibiotics.
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

6. Other Pre Specified Outcome: The Percentage of Subjects With Malignancies (Excluding Carcinoma in Situ of the Cervix).
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

7. Other Pre Specified Outcome: The Percentage of Subjects With Non-melanoma Skin Cancer.
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

8. Other Pre Specified Outcome: The Percentage of Subjects With Major Adverse Cardiovascular Events.
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Percentage of Subjects With Melanoma Skin Cancer.
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The Percentage of Subjects With Injection Site Reactions (eg. Pain, Erythema, Edema Etc)
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: The Percentage of Subjects With Study Treatment Related Hypersensitivity Reactions (eg, Anaphylaxis, Urticaria, Angioedema, Etc).
Description: Primary Safety Endpoint
Time Frame: Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 Weeks
Groups:
- Tildrakizumab 100mg: Subjects received Tildrakizumab 100 mg up to week 16
Arm/Group | Tildrakizumab 100mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 2/51 | 1/48
Other Adverse Events (participants affected / at risk) | 24/51 | 17/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 100mg (N=51) | Placebo (N=48)
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 1 | 0
Ureteric rupture (Renal and urinary disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 100mg (N=51) | Placebo (N=48)
COVID-19 (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Hordeolum (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Chlamydial infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 1
Allergy to chemicals (Immune system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT03897075/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03897075/SAP_001.pdf